CLINICAL TRIAL: NCT00938080
Title: A Phase 1b, Multi-center, Single Blinded, Placebo-controlled, Sequential Dose Escalation Study to Assess the Safety and Tolerability of Topically Applied AG013 in Subjects Receiving Induction Chemotherapy for the Treatment of Cancers of the Head and Neck
Brief Title: Study to Assess Safety and Tolerability of AG013 in Oral Mucositis in Subjects Receiving Induction Chemotherapy for the Treatment of Cancers of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ActoGeniX N.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: AG013-ODOM-101; RAC0810-942
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- AG013: one mouth rinse/day (Experimental)
  Interventions: Biological: AG013
- AG013: three mouth rinses/day (Experimental)
  Interventions: Biological: AG013
- AG013: six mouth rinses/day (Experimental)
  Interventions: Biological: AG013
- one mouth rinse/day (Placebo Comparator)
  Interventions: Other: Placebo
- three mouth rinses/day (Placebo Comparator)
  Interventions: Other: Placebo
- six mouth rinses/day (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AG013 — Mouth rinse once a day for 14 days
  Arms: AG013: one mouth rinse/day
Biological: AG013 — Mouth rinse three times a day for 14 days
  Arms: AG013: three mouth rinses/day
Biological: AG013 — Mouth rinse six times a day for 14 days
  Arms: AG013: six mouth rinses/day
Other: Placebo — Mouth rinse once a day for 14 days
  Arms: one mouth rinse/day
Other: Placebo — Mouth rinse three times a day for 14 days
  Arms: three mouth rinses/day
Other: Placebo — Mouth rinse six times a day for 14 days
  Arms: six mouth rinses/day

SUMMARY:
The purpose of this study is to assess the safety and tolerability of AG013 (genetically modified L. lactis bacteria engineered to secrete human Trefoil Factor 1), and to explore the ability of AG013 to attenuate the course and severity of oral mucositis (OM) in subjects receiving induction chemotherapy for the treatment of head and neck cancer.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety and tolerability of AG013 in subjects who are at risk for oral mucositis (OM) and to assess clinical efficacy of AG013 in the reduction of signs and symptoms of OM in patients receiving induction chemotherapy for the treatment of their head and neck cancer.

AG013 is made up of genetically modified (GM) bacteria called Lactococcus lactis (L. lactis). Wild type L. lactis are commonly used to produce dairy products including cheeses and milk. To make AG013, the DNA of L. lactis has been changed in the laboratory to secrete a protein called human Trefoil Factor 1 (hTFF1). hTFF1 is normally secreted in saliva and intestines. Trefoil factors have been shown to be important in protecting and healing mucosal tissues, such as the tissue in the mouth, when these tissues are damaged by cancer therapies such as chemotherapy and radiation therapy.

The proposed Phase 1b clinical trial will enroll subjects with head and neck cancer who develop OM during their first cycle of treatment with induction chemotherapy. OM is a painful, common toxicity of many forms of drug and radiation therapy used for the treatment of cancer. Subjects with OM get soreness, irritation, and ulcers in the mouth and may have difficulties eating, drinking or swallowing as a result of their cancer treatment.

During the second cycle of induction chemotherapy, eligible subjects will receive AG013 or placebo for 14 consecutive days at a frequency of one rinse, three rinses or six rinses per day (sequential dose escalation design).

At least 21 subjects will be enrolled in the study. For each of the three daily dose levels, 5 subjects will be assigned to AG013 (n=5) and 2 subjects will be assigned to placebo (n=2).

Throughout the study, safety will be monitored by collecting and recording Adverse Events, laboratory assessments and the presence of sAGX0085 bacteria in blood.

An independent Data Safety Monitoring Board (DSMB) will be constituted before the enrollment of subjects in order to review safety data from each enrollment group.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign the study specific Informed Consent Form (ICF) approved by the site's Institutional Review Board
* Males or females 18 years or older
* Recently diagnosed with pathologically-confirmed squamous cell carcinoma of the head and neck (e.g., oral cavity, oropharynx, hypopharynx, larynx, nasopharynx, lips, sinuses, salivary glands, unknown primary)
* Planned to receive at least two cycles of induction chemotherapy of the same regimen consisting of cisplatin/fluorouracil (PF) or cisplatin/fluorouracil/docetaxel (PFT). The planned CT cycles must be of the same length and must be a minimum of 14 days in length
* Karnofsky performance score ≥ 60%
* Screening laboratory assessments:
* Hemoglobin ≥ 10g/dl
* White blood count ≥ 3500 cells/mm3
* Absolute neutrophil counts ≥ 1500 cells/ mm3
* Direct bilirubin ≤ 2x upper limit of normal (ULN)
* Serum AST and ALT ≤ 3 x ULN
* Serum creatinine ≤ 2 mg/dl
* Serum pregnancy test: negative for females of childbearing potential: A women is considered to be of child bearing potential unless she has had a tubal ligation or is postmenopausal (without a menstrual period for at least one year)
* Subjects of childbearing potential must agree to utilize effective contraceptive methods of birth control during study participation and for 30 days following the last treatment with IMP
* Have documented mouth pain during CT Cycle 1 (i.e., OMDQ question 2 score of ≥ 2 during CT Cycle 1)

Exclusion Criteria:

* Prior radiation to the head and neck
* Chemotherapy within 21 days prior to study start
* Presence of active infectious disease excluding oral candidiasis
* Current use of antibiotic rinses or troches
* Alcohol abuse syndrome; recovered alcoholics may be included
* Presence of OM (WHO Grade > 0)
* Chronic immunosuppression
* Known seropositive for HIV or hepatitis B or C
* Use of investigational agent within 30 days of signing informed consent
* Teeth extractions within 7 days prior to the start of CT administration
* Female subjects who are pregnant or nursing
* Known sensitivity to any investigational agent
* Inability to give informed consent or comply with study requirements
* Unwilling or unable to complete subject diary
* Any other clinical condition, psychiatric condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable or to comply with follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse Events, laboratory assessments and the presence of sAGX0085 bacteria in blood) | 16 months
  Up to 16 months

SECONDARY OUTCOMES:
Pharmacokinetics of serum samples, buccal smears and saliva samples | 28 days
  Day 1 CT cycle 2, Day 7 CT cycle 2, Day 14 CT cycle 2, End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Robert S, Steidler L. Recombinant Lactococcus lactis can make the difference in antigen-specific immune tolerance induction, the Type 1 Diabetes case. Microb Cell Fact. 2014 Aug 29;13 Suppl 1(Suppl 1):S11. doi: 10.1186/1475-2859-13-S1-S11. Epub 2014 Aug 29. PMID 25185797